CLINICAL TRIAL: NCT06704464
Title: Investigation of Validity and Reliability of the Minnesota Manual Dexterity Test in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Kader Eldemir, Assistant professor, Cumhuriyet University
Other Study IDs: 1-MS-minnesota-reliability
Record Dates: First submitted 2024-11-18; First posted 2024-11-26 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Minnesota manual dexterity; reliability; validity; multiple sclerosis; hand function
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: Patients with Multiple Sclerosis
  Interventions: Other: Manual Dexterity; Other: disability level
- Control Group: healthy controls
  Interventions: Other: Manual Dexterity (only MMDT)

INTERVENTIONS:
Other: Manual Dexterity — Individuals who meet the inclusion criteria will be evaluated for manual dexterity using MMDT, 9-HPT, ABILHAND, and JTHFT.
  Groups: Test Group
Other: Manual Dexterity (only MMDT) — Individuals who meet the inclusion criteria will be evaluated for manual dexterity using MMDT on a predetermined day.
  Groups: Control Group
Other: disability level — Individuals who meet the inclusion criteria will be evaluated for disability level using EDSS
  Groups: Test Group

SUMMARY:
Many assessment tools have been developed and used to evaluate upper extremity functions in multiple sclerosis (MS) patients. While each test has its strengths and weaknesses, the most significant limitation of these tests is that only a limited number assess both hands simultaneously. On the other hand, most daily life activities require the coordinated use of both hands. In MS patients, bilateral impairments in hand functions can also be observed. Therefore, there is a need for bilateral assessment tools.

Unlike many other assessment tools, the Minnesota Manual Dexterity Test (MMDT) allows for simultaneous evaluation of both hands. In addition to manual dexterity, it also assesses hand-eye coordination and gross motor skills. The MMDT consists of five subtests: placing, turning, displacing, single-hand turning and placing, and two-hand turning and placing. The validity of the MMDT has also been examined in MS patients.

Our study aims to evaluate the reliability and validity of the MMDT in MS patients. The cutoff times that best distinguish individuals with MS from healthy individuals will also be examined. The study aims to systematically and thoroughly evaluate the MMDT, establish it as a valid and reliable method for MS patients, and provide a new perspective on assessing hand functions.

DETAILED DESCRIPTION:
At baseline, the MMDT, EDSS, 9-hole peg test (9-HPT), ABILHAND survey, and Jebsen-Taylor Hand Function Test (JTHFT) will be applied to the MS group. The MMDT will be repeated seven days after the first application in MS. Healthy controls are going to perform only the MMDT.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years,
* Neurologist-diagnosed Multiple Sclerosis,
* Expanded Disability Status Scale (EDSS) score between 0-6.5
* No MS exacerbation within the last 3 months,
* Use of stable medication in the last 3 months.

Exclusion Criteria:

* Having any vision, hearing or perception problems that may affect the research results,
* Having an orthopedic problem that may affect manual skills in the upper extremity,
* Having a cardiovascular, pulmonary disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis who apply to Sivas Cumhuriyet University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Minnesota Manual Dexterity Test | baseline (on the predetermined assessment day)
  The Minnesota Manual Dexterity Test (MMDT) is a performance test designed to evaluate hand functions and hand-eye coordination both unilaterally and bilaterally, higher scores mean a worse outcome.
Minnesota Manual Dexterity Test-second | the second assessment will be conducted after the seven days
  The Minnesota Manual Dexterity Test (MMDT) is a performance test designed to evaluate hand functions and hand-eye coordination both unilaterally and bilaterally, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
9-Hole Peg Test | baseline (on the predetermined assessment day)
  The 9-Hole Peg Test (9-HPT) evaluates hand dexterity based on performance, higher scores mean a worse outcome.
ABILHAND | baseline (on the predetermined assessment day)
  to assess for performance of activity. score range 0-46 point, higher scores mean a better outcome.
The Jebsen Hand Function Test | baseline (on the predetermined assessment day)
  The Jebsen Hand Function Test (JHFT) is one of the objective and standardized tests that assesses fine motor skills and functional hand use by simulating daily living activities, higher scores mean a worse outcome.
The Expanded Disability Status Scale | baseline (on the predetermined assessment day)
  The Expanded Disability Status Scale (EDSS) is a scale used to determine the degree of disability resulting from multiple sclerosis (MS). It evaluates eight functional domains: pyramidal, cerebellar, brainstem, sensory, bowel/bladder, visual, mental, and other functions.Score range 0-10, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet Üniversity, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Celik RGG. Upper Extremity Capability Tests in Multiple Sclerosis. Noro Psikiyatr Ars. 2018;55(Suppl 1):S54-S57. doi: 10.29399/npa.23338. PMID 30692857
- [Result] Hervault M, Balto JM, Hubbard EA, Motl RW. Reliability, precision, and clinically important change of the Nine-Hole Peg Test in individuals with multiple sclerosis. Int J Rehabil Res. 2017 Mar;40(1):91-93. doi: 10.1097/MRR.0000000000000209. PMID 28059944